CLINICAL TRIAL: NCT05270057
Title: A Multicenter Phase 1, Open-Label Trial of Loncastuximab Tesirine in Combination With DA-EPOCH-R in Patients With Previously Untreated Aggressive B-cell Lymphoid Malignancies
Brief Title: Loncastuximab Tesirine in Combination With DA-EPOCH-R in Patients With Previously Untreated Aggressive B-cell Lymphoid Malignancies
Acronym: LONCA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mehdi Hamadani, Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO43132
Record Dates: First submitted 2022-02-24; First posted 2022-03-08 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: B-cell Lymphoma; Burkitt Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma | interventions — Etoposide; etoposide phosphate; Doxorubicin; liposomal doxorubicin; Cyclophosphamide; Rituximab; Vincristine; Prednisone; loncastuximab tesirine

STUDY DESIGN:
Intervention Model Description: Phase 1a will involve a standard 3+3 dose escalation design to find the maximal tolerated dose (MTD) and/or recommended dose for expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Loncastuximab Tesirine Dose Escalation 0.075 mg/kg by IV. (Experimental): The study uses a classic 3+3 dose-escalation design. Three patients will be enrolled into a cohort receiving 0.075 mg/kg by IV. If there is no dose-limiting toxicity (DLT) seen in any of these participants, the trial will enroll additional participants into the next higher dose cohort, which is 0.12 mg/kg by IV. If one patient experiences a DLT at a specific dose, an additional three individuals will be accrued into that same dose cohort. The third dose level is 0.15 mg/kg by IV. DLTs in two or more at a specific dose level indicates that the MTD has been exceeded; dose escalation will not be pursued, and the prior dose level will be expanded to six patients; if there is no more than one patient who experiences a DLT among those six patients, that dose level is considered the MTD.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Prednisone; Drug: Loncastuximab Tesirine 0.075 mg/kg by IV
- Loncastuximab Tesirine Dose Escalation 0.12 mg/kg by IV. (Experimental): The study uses a classic 3+3 dose-escalation design. Three patients will be enrolled into a cohort receiving 0.075 mg/kg by IV. If there is no dose-limiting toxicity (DLT) seen in any of these participants, the trial will enroll additional participants into the next higher dose cohort, which is 0.12 mg/kg by IV. If one patient experiences a DLT at a specific dose, an additional three individuals will be accrued into that same dose cohort. The third dose level is 0.15 mg/kg by IV. DLTs in two or more at a specific dose level indicates that the MTD has been exceeded; dose escalation will not be pursued, and the prior dose level will be expanded to six patients; if there is no more than one patient who experiences a DLT among those six patients, that dose level is considered the MTD.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Prednisone; Drug: Loncastuximab tesirine 0.12 mg/kg by IV
- Loncastuximab Tesirine Dose Escalation 0.15 mg/kg by IV. (Experimental): The study uses a classic 3+3 dose-escalation design. Three patients will be enrolled into a cohort receiving 0.075 mg/kg by IV. If there is no dose-limiting toxicity (DLT) seen in any of these participants, the trial will enroll additional participants into the next higher dose cohort, which is 0.12 mg/kg by IV. If one patient experiences a DLT at a specific dose, an additional three individuals will be accrued into that same dose cohort. The third dose level is 0.15 mg/kg by IV. DLTs in two or more at a specific dose level indicates that the MTD has been exceeded; dose escalation will not be pursued, and the prior dose level will be expanded to six patients; if there is no more than one patient who experiences a DLT among those six patients, that dose level is considered the MTD.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Prednisone; Drug: Loncastuximab tesirine 0.15 mg/kg by IV
- Loncastuximab Tesirine Dose Escalation Maximum Tolerated Dose (Experimental): The study uses a classic 3+3 dose-escalation design. Three patients will be enrolled into a cohort receiving 0.075 mg/kg by IV. If there is no dose-limiting toxicity (DLT) seen in any of these participants, the trial will enroll additional participants into the next higher dose cohort, which is 0.12 mg/kg by IV. If one patient experiences a DLT at a specific dose, an additional three individuals will be accrued into that same dose cohort. The third dose level is 0.15 mg/kg by IV. DLTs in two or more at a specific dose level indicates that the MTD has been exceeded; dose escalation will not be pursued, and the prior dose level will be expanded to six patients; if there is no more than one patient who experiences a DLT among those six patients, that dose level is considered the MTD. This dose will be added to this record when it is determined.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Prednisone; Drug: Loncastuximab Tesirine 0.075 mg/kg by IV; Drug: Loncastuximab tesirine 0.12 mg/kg by IV; Drug: Loncastuximab tesirine 0.15 mg/kg by IV
- Dose Expansion Phase (Experimental): Subjects will receive the recommended phase 2 dose (RP2D) identified from dose-escalation phase. This dose will be added to this record when it is determined.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Vincristine; Drug: Prednisone; Drug: Loncastuximab Tesirine 0.075 mg/kg by IV; Drug: Loncastuximab tesirine 0.12 mg/kg by IV; Drug: Loncastuximab tesirine 0.15 mg/kg by IV

INTERVENTIONS:
Drug: Etoposide — Dose level -2=50 mg/m^2; dose level -1=50 mg/m^2; dose level 1=50 mg/m^2; dose level 2=60 mg/m^2; dose level 3=72 mg/m^2; dose level 4=86.4 mg/m^2; dose level 5=103.7 mg/m^2; dose level 6=124.4 mg/m^2; dose level 7=149.3 mg/m^2
  Other Names: Etopophos; Toposar; Vepesid
Drug: Doxorubicin — Dose level -2=10 mg/m^2; dose level -1; dose level -1=10 mg/m^2; dose level 1=10 mg/m^2; dose level 2=12 mg/m^2; dose level 3=14.4 mg/m^17.3 mg/m^2; dose level 4=17.3 mg/m^2; dose level 5=20.7 mg/m^2; dose level 6=24.8 mg/m^2; dose level 7=29.8 mg/m^2.
  Other Names: Lipodox; Lipodox 50; Doxil; Adriamycin; Rubex
Drug: Cyclophosphamide — Dose level -2=480 mg/m^2; dose -1=600 mg/m^2; dose level 1=750 mg/m^2; level 2=900 mg/m^2; level 3=1080 mg/m^2; level 4=1296 mg/m^2; level 5=1555 mg/m^2; level 6=1866 mg/m^2; level 7=2239 mg/m^2.
  Other Names: Cytoxan; Neosar; Endoxan; Procytox; Revimmune
Drug: Rituximab — Level -2 through level 7: 375 mg/m^2
  Other Names: Rituxan; MabThera
Drug: Vincristine — Level -2 through level 7: 0.4 mg/m^2/day
  Other Names: Oncovin; Vincasar; Marqibo; Leurocristine
Drug: Prednisone — Level -2 through level 7: 60 mg/m^2/twice daily (BID)
  Other Names: Deltasone; Orasone; Meticorten; Liquid Pred
Drug: Loncastuximab Tesirine 0.075 mg/kg by IV — Cohort 1: 0.075 mg/kg by IV. The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: Zynlonta; ADCT-402; loncastuximab tesirine-lpyl
  Arms: Dose Expansion Phase; Loncastuximab Tesirine Dose Escalation 0.075 mg/kg by IV.; Loncastuximab Tesirine Dose Escalation Maximum Tolerated Dose
Drug: Loncastuximab tesirine 0.12 mg/kg by IV — Cohort 2: 0.12 mg/kg by IV. The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: Zynlonta; ADCT-402; loncastuximab tesirine-lpyl
  Arms: Dose Expansion Phase; Loncastuximab Tesirine Dose Escalation 0.12 mg/kg by IV.; Loncastuximab Tesirine Dose Escalation Maximum Tolerated Dose
Drug: Loncastuximab tesirine 0.15 mg/kg by IV — Cohort 3: 0.15 mg/kg by IV The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: Zynlonta; ADCT-402; loncastuximab tesirine-lpyl
  Arms: Dose Expansion Phase; Loncastuximab Tesirine Dose Escalation 0.15 mg/kg by IV.; Loncastuximab Tesirine Dose Escalation Maximum Tolerated Dose

SUMMARY:
The overarching hypothesis for this study is that a safe and tolerable dose (i.e., the maximum tolerated dose) will be identified for loncastuximab tesirine in combination with dose-adjusted etoposide phosphate, prednisone, vincristine sulfate (Oncovin), cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), and rituximab (DA-EPOCH-R) for patients with previously untreated aggressive B-cell lymphoid malignancies.

DETAILED DESCRIPTION:
This is a multicenter phase 1, open-label trial that will evaluate the safety and tolerability of loncastuximab tesirine in combination with DA-EPOCH-R.

Phase 1a will involve a standard 3+3 dose escalation design to find the maximum tolerated dose (MTD) and/or recommended dose for expansion. The MTD will be determined based on the results of the safety evaluation. No intra-patient dose escalation is allowed.

Phase 1b will involve a cohort expansion at the dose level determined to be the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Adult patients with B-cell lymphoma, specifically one of the following: high-grade B-cell lymphoma with MYC and B-cell lymphoma 2 (BCL2) and/or B cell lymphoma 6 (BCL6) rearrangements; high-grade B-cell lymphoma, not otherwise specified, primary mediastinal diffuse large B-cell lymphoma; Burkitt lymphoma; diffuse large B-cell lymphoma with MYC rearrangement; or Cluster of Differentiation 19 (CD19) -positive plasmablastic lymphoma.
3. Patients must not have received prior multiagent chemotherapy for their lymphoma. Limited palliative radiation is allowed. Corticosteroid therapy in symptomatic patients will be permitted and does not require a washout period. Prephase treatment with cyclophosphamide and corticosteroids or vincristine and corticosteroids is allowed in symptomatic patients.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status criteria of 0-3.
5. Adequate hematological function, defined as absolute neutrophil count (ANC) ≥1 × 103/μL and platelet count ≥50 x 10^3/μL.

   - These requirements do not apply to patients with bone marrow involvement of lymphoma.
6. Adequate hepatic function: aspartate aminotransferase (AST) / alanine aminotransferase (ALT) / gamma-glutamyl transferase (GGT) ≤ 3 x institutional upper limit of normal (ULN) and bilirubin < 1.5 x ULN, unless due to hepatic involvement with lymphoma or Gilbert's syndrome.

   - Exceptions can be granted from principal investigator for primarily indirect bilirubinemia if due to recent transfusion and/or hemolysis.
7. Creatinine clearance ≥ 30 ml/min calculated using the Cockroft-Gault formula.
8. Left ventricular ejection fraction (LVEF) of ≥50%, assessed by echocardiography or cardiac multi-gated acquisition (MUGA) scan.
9. Patients with marrow-only disease will be eligible.
10. Patients rendered no evidence of disease via surgery will be eligible.
11. Central nervous system (CNS) involvement is not considered contraindication for patients with Burkitt lymphoma.
12. Known HIV-positive patients compliant with antiretroviral therapy and with undetectable viral loads will be permitted.
13. Pregnancy It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below.

    * Female patients of childbearing potential must use a highly effective method of contraception during the entire study treatment period and through nine months after the last dose of loncastuximab tesirine.
    * Male patients, even if surgically sterilized (i.e., status postvasectomy), with female partners who are of childbearing potential should use a condom when sexually active during the entire study treatment period and through six months after the last dose of loncastuximab tesirine.
14. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Presence of clinically significant pericardial or pleural effusions, or third space fluid accumulations (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
2. Known history of hypersensitivity to CD19 antibody, components of study medication, or DA-EPOCH-R.
3. Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy. These subjects MUST HAVE undetectable HBV viral load to be considered for this protocol.
4. Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load.
5. Breastfeeding or pregnant.
6. Active systemic bacterial, viral, fungal, or other infection requiring systemic treatment at time of screening.
7. Congenital long QT syndrome or a corrected QT measure (QTc) interval of >480 ms at screening (unless secondary to pacemaker or bundle branch block).
8. Patients diagnosed with another malignancy within three years or with any evidence of residual prior malignant disease (except nonmelanoma skin cancer, non-metastatic prostate cancer, in situ cervical cancer, or ductal or lobular carcinoma in situ). Patients meeting this exclusion criteria may be enrolled after approval from study PI.
9. Significant medical comorbidities such as New York Heart Association class ≥III heart failure, unstable angina, uncontrolled arrhythmias, or severe chronic pulmonary disease.
10. Lymphoma with active CNS involvement at time of screening unless the patient has Burkitt lymphoma.
11. Patient with known intraparenchymal CNS involvement (including those with Burkitt lymphoma).
12. Patients with known Child Pugh Class C hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD). | Up to 21 days (one cycle) for each dosing cohort.
  MTD is defined as the highest dose level where zero of the first three patients treated or ≤1 of the first six patients treated had a dose-limiting toxicity (DLT) during cycle 1 of phase 1a.
The number of dose-limiting toxicities (dose-escalation phase only). | Up to 21 days (one cycle).
  A dose-limiting toxicity is defined as any of the following within 21 days after administration of the first dose of loncastuximab tesirine in phase 1a part 1a only (except any toxicity clearly due to disease or other causes): adverse events and lab data, using Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hamadani, MD, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - University of Texas Southwestern, Dallas, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No